CLINICAL TRIAL: NCT06379932
Title: Exploring Pain: Prospective Observational Study on Pain Perception During and After Muscle Biopsy
Brief Title: Pain and Muscle Biopsy
Acronym: BIODOMU
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP240433
Record Dates: First submitted 2024-04-18; First posted 2024-04-23 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Neuromuscular Diseases
Keywords: pain; neuromuscular disease; open muscle biopsy
MeSH Terms: conditions — Neuromuscular Diseases; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Surveys completion — A questionnaire (including the NRS) will be given to the patient on the day of the procedure, immediately after the biopsy, in the treatment room and without staff intervention (responses will be analyzed by two study investigators at a later date).
  The patient health questionnaire (PHQ-9) will also be provided at the same time as the self-report questionnaire, for the assessment of depressive symptoms.
  Assessment of the participant's frailty using the Clinical Frailty Scale (CFS) will be carried out prior to the procedure.
  Further data will be collected by telephone by a study investigator 15 +/- 2 days after the biopsy and 30 +/- 2 days after the biopsy.

SUMMARY:
Few studies have been conducted on pain assessment during and after open muscle biopsy. Furthermore, no clinical factors likely to influence pain perception during and after open muscle biopsy have been evaluated in previous studies.The proposed observational study aims to study pain perception in subjects over the aged of 18 years old who underwent an open muscle biopsy for a suspected myopathic disorder. Describing the main characteristics of pain during and after open muscle biopsy using a questionnaire will not only clarify this aspect, which is little studied in the literature, but will also provide information for improving analgesic management of the procedure.Studying the prognostic aspects of pain perception will give healthcare professionals an idea of which patients are at risk of suffering greater adverse effects from the procedure, so that they can be offered a personalised service in the future.

DETAILED DESCRIPTION:
The patients will be followed for 30 days +/-2 days from the date of inclusion (day de la biopsy). The duration of the inclusion period will be 5 months. The total duration of the study until the phone call to the last patient included will be 6 months +/- 2 days.Sample size estimated: 100 patients, both male and female. Patients will present to the study site for a scheduled diagnostic muscle biopsy, with no additional visits required for study data collection. Prior to performing the procedure as part of the care, the investigator will verify that the inclusion and non-inclusion criteria are met and the patient will be informed of the opportunity to participate in this study. The study investigator will explain the details of the study (including the objective and how it will be carried out) and will obtain the patient's non-opposition to the study. Assessment of the participant's frailty using the frailty scale will be carried out prior to the procedure as part of the care.

The overall assessment of the patient on the day of the procedure will be carried out in accordance with the standard of care and will include the collection of vital signs parameters, height and weight.

The biopsy will be carried out in accordance with the department's care protocol. The self-reported questionnaire assessing pain during and after muscle biopsy (investigator-generated) and including NRS (Numerical Rating Scale) will be provided on the day of the procedure, immediately after the biopsy, in the treatment room and without staff intervention (responses will be analysed by two study physicians at a later date). The patient health questionnaire (PHQ-9) will also be provided at the same time as the self-report questionnaire for the assessment of depressive symptoms. Other data will be collected by telephone by a study investigator 15 days +/- 2 days after the biopsy and 30 days +/- 2 days after the biopsy. Responses will be analysed pseudonymously and will not prejudge the patient's continued treatment.Once collected, the paper data is organised, cleaned and stored appropriately in the paper CRF and transferred to Excel. Data obtained during telephone interviews will be entered directly into the Excel CRF. Medical data from the medical records will be transferred to Excel.

Two study investigators will enter and validate the data, including data quality control measures to ensure accuracy and reliability.

The data collected will be analysed by the investigators using the following statistical methods: descriptive statistics to summarise the characteristics of the study population and inferential statistics to test hypotheses or associations between variables. After analysing the data, the researchers interpret the results in the context of the research question and the existing literature. "

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years
* Patients with clinical suspicion of myopathy.
* Patients requiring open muscle biopsy in the neuropathology unit at GH Pitié Salpêtrière.
* Patients who do not object to their participation in the study."

Exclusion Criteria:

* Patients who do not understand French.
* Pregnant women
* No social security and patient under AME.
* Patient deprived of liberty by court or administrative order, or under legal protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adults undergoing open muscle biopsy for suspicion of neuromuscular disorder
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2024-08-06 (Actual); Primary Completion 2025-06-12 (Actual); Study Completion 2025-06-12 (Actual)

PRIMARY OUTCOMES:
To describe the characteristics and intensity of pain during and after open muscle biopsy on the basis of a questionnaire including NRS scale. | Day of musclebiopsy until 30 days +/- 2 days after the biopsy
  Completion of a questionnaire after the biopsy. The questionnaire is made up of several sections of questions, which will assess preoperative aspects (anxiety, quality of information received from healthcare staff) and intraoperative aspects, such as the assessment of perceived pain using the NRS scale. The questionnaire, which lasts around 5-10 minutes, is completed by the patient independently.
  Information on post-operative progress will be gathered during two follow-up telephone interviews at 15 and 30 days. These interviews will consist of answering the questions in the second part of the questionnaire and will last approximately 10 minutes.

SECONDARY OUTCOMES:
To identify prognostic factors that may influence pain perception and to gather opinions to improve quality service | Day of musclebiopsy until 30 days +/- 2 days after the biopsy
  The following elements will be evaluated: personal information (age, sex, patient already treated for chronic pain), result of the PHQ9 questionnaire validated for the evaluation of depressive symptoms, Frailty scale and response to the self-declared questionnaire (preoperative anxiety) including the NRS. The PHQ9 questionnaire will be given at the same time as the pain assessment questionnaire, after the biopsy. The frailty scale will be carried out by the investigator at the time of the pre-biopsy clinical assessment.
  All the above variables will be correlated with the data obtained from the self-report questionnaire (numerical pain rating scale - NRS) and the telephone interviews (use of analgesics during follow-up).
Gather patient feedback on procedures, facilities and reception to improve our service to patients. | Day of musclebiopsy
  Assessment of possible measures to improve our services to patients, based on analysis of patient comments and responses to sections 1 to 7 of the self-declared questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Teresinha Maria DIAS EVANGELISTA, Principal Investigator — Sorbonne University, Pitié salpêtrière hospital
Locations (1):
- Pitié-Salpêtrière, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients. Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal